CLINICAL TRIAL: NCT02756832
Title: Local, Multicentre, Observational, Non-Interventional Prospective Study of Alogliptin Benzoate in Patients With Diabetes Mellitus Type 2
Brief Title: An Observational Study of Alogliptin Benzoate in Participants With Diabetes Mellitus Type 2
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Alogliptin-4018; MACS-2015-101024 (Other: Takeda)
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alogliptin Benzoate: Participants with diabetes mellitus type 2 (T2DM) who received alogliptin benzoate tablets, orally, as prescribed by physician according to Russian summary of product characteristics (SmPC) were observed for approximately 6 months.
  Interventions: Drug: Alogliptin Benzoate

INTERVENTIONS:
Drug: Alogliptin Benzoate — Alogliptin benzoate tablets
  Other Names: VIPIDIA®

SUMMARY:
The purpose of this study is to evaluate the effect of alogliptin benzoate (VIPIDIA®) on glycosylated hemoglobin (HbA1c) level dynamics in participants with diabetes mellitus type 2 (T2DM) at Month 6.

DETAILED DESCRIPTION:
The drug being studied in this study is called alogliptin benzoate. Alogliptin benzoate is being researched to treat people who have T2DM. This study will look at the HbA1c level dynamics in participants with T2DM.

The study enrolled 1409 patients. Alogliptin benzoate will be prescribed by their physician in accordance with the Russian summary of product characteristics (SmPC).

This multi-center study will be conducted in the Russian Federation. The overall duration of study for observation will be approximately 6 months. Participants will make multiple visits to the clinic as assigned by each physician according to their routine practice, in every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥ 18 years of age;
2. Has a diagnosis of type 2 diabetes mellitus (T2DM)
3. Participants with:

   * newly diagnosed diabetes mellitus (DM) type 2 (drug naïve) or
   * inadequate glycemic control on previously prescribed any oral antidiabetic drug.
4. VIPIDIA® is prescribed according to the approved label for the Russian Federation.
5. The participant's physician decides to prescribe VIPIDIA®:

   * as monotherapy or
   * as a part of combination therapy.
6. The participant (or, when applicable, the participant's legally acceptable representative) signs and dates a written, informed consent form prior to the start of data collection. Participant is capable of understanding the written informed consent, provides signed and written informed consent, and agrees to comply with protocol requirements. In case the participant is blind or unable to read, informed consent will also be witnessed.

Exclusion Criteria:

1. Contraindications of respective approved Russian summary of product characteristics (SmPC);
2. In the opinion of the physician, the participant has any reasons of medical and non-medical character, which in the opinion of the physician can prevent participant participation in the study;
3. Had used Dipeptidyl peptidase-4 inhibitors (DPP-IV inhibitors) or Glucagon like peptide-1 agonists (aGLP-1) within the 3 months prior to the start of VIPIDIA® treatment.
4. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with type 2 diabetes mellitus (T2DM) will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 1409 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (52):
- Russia (52):
  - First City Clinical Hospital named after E.E. Vlosevich, Arkhangelsk
  - City polyclinic #11, Barnaul
  - Belgorod Regional Clinical hospital named after Saint I Belgorod Regional Clinical Hospital of St. Joasaph, Belgorod
  - LLC Medical center Lotos, Chelyabinsk
  - Istochnik clinic, Chelyabinsk
  - Regional clinical hospital #3, Chelyabinsk
  - Medical center Health Academy, Chita
  - Chita State Medical Academy, Chita
  - City polyclinic #11, Kazan'
  - Ciry polyclinic #10, Kazan'
  - Kemerovo Regional Clinical Hospital named after S.V. Belyaev, Kemerovo
  - Medical Center Clinic of Hormonal Health, Khabarovsk
  - Regional Clinical hospital named after S.I. Sergeev, Khabarovsk
  - Road Clinical Hospital at Khabarovsk Station - 1, Khabarovsk
  - Northern Clinical Emergency Hospital, Kirov
  - Kirov Clinical Hospital #7 named after V.I. Yurlova, Kirov
  - Kostroma City hospital, Kostroma
  - Kursk Regional Clinical Hospital, Kursk
  - Lobnya Central City Hospital, Lobnya
  - City polyclinic #166, Moscow
  - Endocrinology Research Center, Moscow
  - City polyclinic #22, Moscow
  - City polyclinic #52, Moscow
  - The Scientific Center of Cardiovascular Surgery named after A.N. Bakulev, Moscow
  - CJSC Medsi, Moscow
  - Diagnostical Center #5, Moscow
  - Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation, Moscow
  - Clinical Diagnostical Center, Nizhny Novgorod
  - City polyclinic #3, Nizhny Novgorod
  - Medical Center Healthy family LLC, Novosibirsk
  - Republican Hospital named after V.A.Baranov, Petrozavodsk
  - Rostov State Medical University, Rostov-on-Don
  - City Clinical hospital #11, Ryazan
  - City policlinic #117, Saint Petersburg
  - City polyclinic #109, Saint Petersburg
  - Saint-Petersburg Territorial Diabetological Center, Saint Petersburg
  - City policlinic #86, Saint Petersburg
  - Consultative and diagnostic polyclinic 1 of Primorsky district, Saint Petersburg
  - Samara Regional Clinical Diagnostical polyclinic #14, Samara
  - LLC Center Diabet, Samara
  - City policlinic #9, Samara
  - City polyclinic #22, Saratov
  - City policlinic #3, Tomsk
  - LLC Medical center Ideale, Tomsk
  - Tomsk Regional Clinical Hospital, Tomsk
  - City polyclinic #43, Ufa
  - Regional Clinical Hospital, Vladimir
  - Regional Clinical Hospital #1, Volgograd
  - Volgograd State Medical University, Volgograd
  - LLC Zdorovye, Diabetes Center, Vologda
  - Voronezh Regional Clinical Diagnostical center, Voronezh
  - Ural State Medical Academy, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study in Russia from 20-Sep-2016 to 28-Apr-2018.
Pre-assignment Details: Participants with a diagnosis of diabetes mellitus type 2 (T2DM) prescribed alogliptin benzoate in accordance with Russian SmPC were enrolled in this observational study.
Period: Overall Study
Arm/Group | Alogliptin Benzoate
Started | 1409
Received Therapy | 1393
Included in Efficacy and Safety Analysis | 1399
Completed | 1356
Not Completed | 53
Not completed — Lost for Observation after Baseline | 6
Not completed — Lost for Observation | 13
Not completed — Patient's Unwillingness | 12
Not completed — Insufficient Efficacy | 2
Not completed — Sponsor Decision/Regulatory Requirement | 1
Not completed — Reason not Specified | 9
Not completed — Protocol Deviation | 10

BASELINE CHARACTERISTICS:
Population: All participants with a diagnosis of diabetes mellitus type 2 (T2DM), newly diagnosed T2DM (drug naive) or inadequate glycemic control on previously prescribed any oral antidiabetic drug were enrolled in the study.
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 907
  Male | 492
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  European | 1375
  Asian | 21
  African American or African | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 1399

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) Level at Month 6
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Month 6 relative to baseline. Glycosylated hemoglobin (HbA1c) as a diagnostic criteria of diabetes mellitus is ≥6.5%. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 6
Population: All participants with a diagnosis of diabetes mellitus type 2 (T2DM), newly diagnosed T2DM (drug naive) or inadequate glycemic control on previously prescribed any oral antidiabetic drug were enrolled in the study. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
percentage of glycosylated hemoglobin
  Baseline: number analyzed (Participants) | 1392
  Baseline | 8.1 (1.2)
  Change from Baseline at Month 6: number analyzed (Participants) | 1314
  Change from Baseline at Month 6 | -1.2 (1.0)

2. Secondary Outcome: Change From Baseline in HbA1c Level at Month 6 in Subgroups of Participants With Different Clinical Characteristics
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Month 6 relative to baseline. Glycosylated hemoglobin (HbA1c) as a diagnostic criteria of diabetes mellitus is ≥6.5%. Subgroups included participants with different baseline clinical characteristics with predictors such as prior therapy of diabetes mellitus, sex, age group, cardiovascular risk group, therapy type (monotherapy or combined therapy), baseline body mass index (BMI) and initial glycemic control and T2DM duration. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 6
Population: All participants with a diagnosis of T2DM, newly diagnosed T2DM (drug naive) or inadequate glycemic control on previously prescribed any oral antidiabetic drug were enrolled in the study. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1314
percentage of glycosylated hemoglobin
  Prior Therapy Diabetes Mellitus (DM), No Therapy: number analyzed (Participants) | 332
  Prior Therapy Diabetes Mellitus (DM), No Therapy | -1.4 (1.2)
  Prior Therapy DM, Monotherapy: Biguanides: number analyzed (Participants) | 629
  Prior Therapy DM, Monotherapy: Biguanides | -1.1 (0.8)
  Prior Therapy DM, Monotherapy: Sulfonylureas: number analyzed (Participants) | 75
  Prior Therapy DM, Monotherapy: Sulfonylureas | -1.3 (1.3)
  Prior Therapy DM, Monotherapy: Other: number analyzed (Participants) | 1
  Prior Therapy DM, Monotherapy: Other | -1.1 (0.0)
  Prior Therapy DM, Biguanides+Sulfonylureas: number analyzed (Participants) | 260
  Prior Therapy DM, Biguanides+Sulfonylureas | -1.3 (1.1)
  Prior Therapy DM, Biguanides+SGLT2 inhibitors: number analyzed (Participants) | 11
  Prior Therapy DM, Biguanides+SGLT2 inhibitors | -1.4 (1.1)
  Prior Therapy DM, Combined therapy: Other: number analyzed (Participants) | 6
  Prior Therapy DM, Combined therapy: Other | -1.8 (1.4)
  Sex, Male: number analyzed (Participants) | 463
  Sex, Male | -1.4 (1.1)
  Sex,Female: number analyzed (Participants) | 851
  Sex,Female | -1.1 (0.9)
  Age Group, <58 Years: number analyzed (Participants) | 588
  Age Group, <58 Years | -1.3 (1.0)
  Age Group, ≥58 Years: number analyzed (Participants) | 726
  Age Group, ≥58 Years | -1.1 (1.0)
  Cardiovascular (CV) Risk Group, High CV Risk: number analyzed (Participants) | 175
  Cardiovascular (CV) Risk Group, High CV Risk | -1.3 (1.1)
  CV Risk Group, Very High CV Risk: number analyzed (Participants) | 1139
  CV Risk Group, Very High CV Risk | -1.2 (1.0)
  Therapy Type (TT), Monotherapy: VIPIDIA®: number analyzed (Participants) | 214
  Therapy Type (TT), Monotherapy: VIPIDIA® | -1.3 (1.1)
  TT, Combined: VIPIDIA®+Biguanides: number analyzed (Participants) | 767
  TT, Combined: VIPIDIA®+Biguanides | -1.1 (0.9)
  TT, Combined: VIPIDIA®+Sulfonylureas: number analyzed (Participants) | 59
  TT, Combined: VIPIDIA®+Sulfonylureas | -1 (1.1)
  TT, Combined: VIPIDIA®+SGLT2 Inhibitors: number analyzed (Participants) | 1
  TT, Combined: VIPIDIA®+SGLT2 Inhibitors | 0 (0)
  TT, Combined: VIPIDIA®+Biguanides+Sulfonylureas: number analyzed (Participants) | 259
  TT, Combined: VIPIDIA®+Biguanides+Sulfonylureas | -1.4 (1.2)
  TT, Combined: VIPIDIA®+Biguanides+SGLT2 Inhibitors: number analyzed (Participants) | 10
  TT, Combined: VIPIDIA®+Biguanides+SGLT2 Inhibitors | -1.3 (1.0)
  TT, Combined: VIPIDIA®+Biguanides+Antidiabetics: number analyzed (Participants) | 1
  TT, Combined: VIPIDIA®+Biguanides+Antidiabetics | -2.4 (0.0)
  TT,Combined: VIPIDIA®+Biguanide+Sulfonylurea+SGLT2: number analyzed (Participants) | 3
  TT,Combined: VIPIDIA®+Biguanide+Sulfonylurea+SGLT2 | -2.1 (0.5)
  BMI, Normal Weight (<25 kg/m^2): number analyzed (Participants) | 72
  BMI, Normal Weight (<25 kg/m^2) | -1.3 (1.2)
  BMI, Over-Weight (25≤BMI<30 kg/m^2): number analyzed (Participants) | 375
  BMI, Over-Weight (25≤BMI<30 kg/m^2) | -1.2 (0.9)
  BMI, Obesity Class I (30≤BMI<35 kg/m^2): number analyzed (Participants) | 502
  BMI, Obesity Class I (30≤BMI<35 kg/m^2) | -1.2 (1.0)
  BMI, Obesity Class II (35≤BMI<40 kg/m^2): number analyzed (Participants) | 259
  BMI, Obesity Class II (35≤BMI<40 kg/m^2) | -1.2 (1.1)
  BMI, Obesity Class III (BMI≥40 kg/m^2): number analyzed (Participants) | 104
  BMI, Obesity Class III (BMI≥40 kg/m^2) | -1.2 (1.2)
  Glycemic Control, HBA1C<7.5%: number analyzed (Participants) | 358
  Glycemic Control, HBA1C<7.5% | -0.6 (0.5)
  Glycemic Control, 7.5%≥HBA1C<9%: number analyzed (Participants) | 713
  Glycemic Control, 7.5%≥HBA1C<9% | -1.1 (0.6)
  Glycemic Control, HBA1C≥9%: number analyzed (Participants) | 243
  Glycemic Control, HBA1C≥9% | -2.5 (1.4)
  T2DM Duration, 0-3 Years: number analyzed (Participants) | 697
  T2DM Duration, 0-3 Years | -1.3 (1.0)
  T2DM Duration, 3-5 Years: number analyzed (Participants) | 133
  T2DM Duration, 3-5 Years | -1.0 (0.9)
  T2DM Duration, 5-10 Years: number analyzed (Participants) | 292
  T2DM Duration, 5-10 Years | -1.2 (0.9)
  T2DM Duration, >=10 Years: number analyzed (Participants) | 190
  T2DM Duration, >=10 Years | -1.2 (1.2)

3. Secondary Outcome: Percentage of Participants With a Decrease in HbA1c Level by <7.0% at Month 6
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Month 6 relative to baseline. Percentage of participants with a decrease of <7.0% from baseline in HbA1c were reported.
Time Frame: Baseline and Month 6
Population: All participants with a diagnosis of T2DM, newly diagnosed T2DM (drug naive) or inadequate glycemic control on previously prescribed any oral antidiabetic drug were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
percentage of participants | 52 [49.2 to 54.7]

4. Secondary Outcome: Change From Baseline in HbA1c Level Over Time
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Months 3 and 6 relative to baseline. Glycosylated hemoglobin (HbA1c) as a diagnostic criteria of diabetes mellitus is ≥6.5%. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
percentage of glycosylated hemoglobin
  Baseline: number analyzed (Participants) | 1392
  Baseline | 8.1 (1.2)
  Change from Baseline to Month 3: number analyzed (Participants) | 1250
  Change from Baseline to Month 3 | -0.8 (0.9)
  Change from Month 3 to Month 6: number analyzed (Participants) | 1220
  Change from Month 3 to Month 6 | -0.4 (0.5)

5. Secondary Outcome: Percentage of Participants With Marked Hyperglycemia at Month 3
Description: Marked hyperglycemia is defined as fasting plasma glucose (FPG) higher than or equal to 11 mmol/L.
Time Frame: Month 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
percentage of participants | 0.9 [0.5 to 1.6]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) Levels Over Time
Description: The change in the value of fasting plasma glucose value collected at Months 3 and 6 relative to baseline. Target FPG depended on the defined individual targets of glycemic control by HbA1c level ≤6.5 to 8.0 mmol/l. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
mmol/l
  Baseline: number analyzed (Participants) | 1323
  Baseline | 8.7 (2.1)
  Change from Baseline to Month 3: number analyzed (Participants) | 1237
  Change from Baseline to Month 3 | -1.7 (1.8)
  Change from Month 3 to Month 6: number analyzed (Participants) | 1225
  Change from Month 3 to Month 6 | -0.4 (0.9)
  Change from Baseline to Month 6: number analyzed (Participants) | 1255
  Change from Baseline to Month 6 | -2.1 (2.0)

7. Secondary Outcome: Change From Baseline in Weight Over Time
Description: Change in the participant's weight was collected at Months 3 and 6 relative to baseline.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
kg
  Baseline: number analyzed (Participants) | 1395
  Baseline | 90.6 (16.5)
  Change from Baseline to Month 3: number analyzed (Participants) | 1377
  Change from Baseline to Month 3 | -1.5 (3.0)
  Change from Month 3 to Month 6: number analyzed (Participants) | 1353
  Change from Month 3 to Month 6 | -1.1 (2.9)
  Change from Baseline to Month 6: number analyzed (Participants) | 1355
  Change from Baseline to Month 6 | -2.6 (4.2)

8. Secondary Outcome: Change From Baseline in Postprandial Glycemia Over Time
Description: The change between the baseline (pre-prandial (before meal)) and postprandial (after meal) glucose values were collected at Months 3 and 6 relative to baseline.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
mmol/l
  Baseline: number analyzed (Participants) | 991
  Baseline | 10.4 (2.2)
  Change from Baseline to Month 3: number analyzed (Participants) | 913
  Change from Baseline to Month 3 | -1.9 (2.0)
  Change from Month 3 to Month 6: number analyzed (Participants) | 989
  Change from Month 3 to Month 6 | -0.5 (1.0)
  Change from Baseline to Month 6: number analyzed (Participants) | 915
  Change from Baseline to Month 6 | -2.4 (2.2)

9. Secondary Outcome: Change From Baseline in Total Cholesterol, Triglycerides, Low Density Lipoproteins and High Density Lipoproteins Over Time
Description: The change between the total cholesterol triglycerides, low density lipoproteins and high density lipoproteins values were collected at Months 3 and 6 relative to baseline.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
mmol/l
  Total Cholesterol, Baseline: number analyzed (Participants) | 1185
  Total Cholesterol, Baseline | 5.6 (1.2)
  Total Cholesterol, Change from Baseline to Month 3: number analyzed (Participants) | 849
  Total Cholesterol, Change from Baseline to Month 3 | -0.5 (0.8)
  Total Cholesterol, Change from Month 3 to Month 6: number analyzed (Participants) | 851
  Total Cholesterol, Change from Month 3 to Month 6 | -0.2 (0.6)
  Total Cholesterol, Change from Baseline to Month 6: number analyzed (Participants) | 967
  Total Cholesterol, Change from Baseline to Month 6 | -0.6 (1.0)
  Triglycerides, Baseline: number analyzed (Participants) | 825
  Triglycerides, Baseline | 2.2 (2.2)
  Triglycerides, Change from Baseline to Month 3: number analyzed (Participants) | 556
  Triglycerides, Change from Baseline to Month 3 | -0.4 (1.7)
  Triglycerides, Change from Month 3 to Month 6: number analyzed (Participants) | 613
  Triglycerides, Change from Month 3 to Month 6 | -0.1 (0.5)
  Triglycerides, Change from Baseline to Month 6: number analyzed (Participants) | 630
  Triglycerides, Change from Baseline to Month 6 | -0.4 (1.6)
  Low Density Lipoproteins (LDL), Baseline: number analyzed (Participants) | 715
  Low Density Lipoproteins (LDL), Baseline | 3.4 (1.1)
  LDL, Change from Baseline to Month 3: number analyzed (Participants) | 433
  LDL, Change from Baseline to Month 3 | -0.4 (0.7)
  LDL, Change from Month 3 to Month 6: number analyzed (Participants) | 482
  LDL, Change from Month 3 to Month 6 | -0.2 (0.6)
  LDL, Change from Baseline to Month 6: number analyzed (Participants) | 525
  LDL, Change from Baseline to Month 6 | -0.6 (0.9)
  High Density Lipoproteins (HDL), Baseline: number analyzed (Participants) | 666
  High Density Lipoproteins (HDL), Baseline | 1.3 (0.5)
  HDL, Change from Baseline to Month 3: number analyzed (Participants) | 396
  HDL, Change from Baseline to Month 3 | 0.0 (0.3)
  HDL, Change from Month 3 to Month 6: number analyzed (Participants) | 441
  HDL, Change from Month 3 to Month 6 | 0.0 (0.3)
  HDL, Change from Baseline to Month 6: number analyzed (Participants) | 473
  HDL, Change from Baseline to Month 6 | 0.1 (0.4)

10. Secondary Outcome: Percentage of Participants With a Decrease in HbA1c Level by ≥0.3% at Month 6
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Month 6 relative to baseline. Percentage of participants with a decrease of ≥0.3% from baseline in HbA1c were reported.
Time Frame: Baseline and Month 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
percentage of participants | 89.1 [87.3 to 90.8]

11. Secondary Outcome: Percentage of Participants Who Used Healthcare Resources
Description: Healthcare resources included rate of hospitalization, emergency, emergency room visits, physician office visits, and other type of usage.
Time Frame: Baseline up to Month 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alogliptin Benzoate
Number analyzed (Participants) | 1399
percentage of participants
  Rate of Hospitalization | 0.6 [0.3 to 1.1]
  Rate of Emergency | 0.1 [0.0 to 0.5]
  Rate of Physician Office Visits | 0.6 [0.3 to 1.1]
  Rate of Other Type of Usage | 0.1 [0.0 to 0.4]

ADVERSE EVENTS:
Time Frame: From first dose of study drug administration up to Month 6
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin Benzoate
All-Cause Mortality (participants affected / at risk) | 0/1399
Serious Adverse Events (participants affected / at risk) | 5/1399
Other Adverse Events (participants affected / at risk) | 69/1399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin Benzoate (N=1399)
Vertebrobasilar insufficiency (Nervous system disorders) | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Schizophrenia (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin Benzoate (N=1399)
Blood cholesterol increased (Investigations) | 10
HbA1C increased (Investigations) | 10
Blood triglycerides increased (Investigations) | 9
Blood glucose increased (Investigations) | 7
Low density lipoprotein increased (Investigations) | 6
High density lipoprotein decrease (Investigations) | 2
Blood creatine increased (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 1
Hypertension (Vascular disorders) | 10
Upper respiratory tract infection (Infections and infestations) | 6
Pyelonephritis chronic (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 2
Viral tracheitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Drug ineffective (General disorders) | 4
Autonomic neuropathy (Nervous system disorders) | 2
Goitre (Endocrine disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Diabetic retinopathy (Eye disorders) | 1
Disease risk factor (Social circumstances) | 1
Vestibular disorder (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT02756832/SAP_000.pdf
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT02756832/Prot_001.pdf